CLINICAL TRIAL: NCT06638671
Title: Short-Term Metformin Use in Young, Healthy Adults: Impacts on the Blood Lactate Response to Exercise and Time-to-exhaustion in a Placebo-controlled, Crossover Study
Brief Title: Short-Term Metformin Use in Young, Healthy Adults: Impacts on Exercise Capacity
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: University of Virginia (Other)
Responsible Party: Principal Investigator, Jason Allen, Associate Professor, University of Virginia
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: HSR240014
Record Dates: First submitted 2024-09-23; First posted 2024-10-15 (Actual); Last update posted 2025-12-18 (Actual); Status verified 2025-12

CONDITIONS: Exercise Capacity; Metformin
Keywords: Exercise capacity; Metformin; Lactate threshold
MeSH Terms: interventions — Metformin

STUDY DESIGN:
Intervention Model Description: Randomized, double-blind, placebo-controlled crossover design
Who Masked: Participant, Investigator
Masking Description: Double-blind
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Metformin (MET) (Experimental): At the end of the screening visit, participants will be randomized to either Condition A or Condition B (MET or PL first). Participants will begin the 19-day treatment phase of study the day after screening.
  During each treatment phase, participants will consume metformin as follows: 1x500 mg tablet/day for 5 days, 2x500 mg tablets/day for 5 days, and 3x500 mg tablets/day (or maximally tolerated dosage) for 9 days.
  Participants will then complete a VO2peak/LT test on day 16, rest for 48 hours, then complete a time-to-exhaustion test (day 19) during the final days of the treatment phase. After the time-to-exhaustion test, participants will begin the placebo treatment phase.
  Interventions: Drug: Metformin Hydrochloride
- Placebo (PL) (Placebo Comparator): At the end of the screening visit, participants will be randomized to either Condition A or Condition B (MET or PL first). Participants will begin the 19-day treatment phase of study the day after screening.
  During each treatment phase, participants will consume placebo as follows: 1x500 mg tablet/day for 5 days, 2x500 mg tablets/day for 5 days, and 3x500 mg tablets/day (or maximally tolerated dosage) for 9 days.
  Participants will then complete a VO2peak/LT test on day 16, rest for 48 hours, then complete a time-to-exhaustion test (day 19) during the final days of the treatment phase. After the time-to-exhaustion test, participants will begin the metformin treatment phase.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Metformin Hydrochloride — Participants will consume metformin or placebo in a randomized order. Participants will complete exercise visits during each treatment phase.
  Arms: Metformin (MET)
Drug: Placebo — Participants will consume metformin or placebo in a randomized order. Participants will complete exercise visits during each treatment phase.
  Arms: Placebo (PL)

SUMMARY:
Metformin is the most prescribed blood sugar (glucose)-lowering medication for patients diagnosed with type 2 diabetes mellitus (T2DM). Metformin stimulates glucose uptake in skeletal muscle similar to the effects of exercise, though, some studies report that metformin may decrease exercise capacity.

The main question this study looks to answer is:

• Does metformin alter exercise capacity?

Participants will:

* Complete 5 exercise tests on a stationary bike.
* Undergo a body composition test.
* Take metformin and placebo.
* Complete food and symptom logs.

The researchers hypothesize that:

• Metformin will reduce aerobic capacity.

DETAILED DESCRIPTION:
Metformin, a potent biguanide, is the most prescribed glucose-lowering medication for patients newly diagnosed with type 2 diabetes mellitus (T2DM). Metformin has purported utility for various conditions such as aging, autoimmune conditions, and cancer, however, the primary use of metformin is for blood glucose reduction via decreased glucose production in the liver (increased glycogenesis, decreased glycogenolysis and gluconeogenesis), reduced glucose absorption in the gut, and enhanced insulin-independent skeletal muscle glucose uptake. The effect of metformin within skeletal muscle is the focus of this study.

The mechanism for improved metformin-mediated skeletal muscle glucose uptake involves the inhibition of complex 1 (NADH:ubiquinone oxidoreductase) in the mitochondrial electron transport chain (ETC). This leads to a reduced cellular energy charge, marked by a reduced ATP concentration and increased ratios of ADP:ATP and AMP:ATP. This energetic imbalance initiates phosphorylation of 5' adenosine monophosphate-activated protein kinase (AMPK), which in turn induces glucose transporter (GLUT4) translocation to the cell membrane and upregulates insulin-independent glucose uptake by skeletal muscle fibers. This cellular energy imbalance and subsequent AMPK signaling cascade is similar to stress elicited by exercise. However, during exercise, the energy imbalance is created by increased ATP utilization from skeletal muscle contraction rather than incomplete glucose metabolism (less ATP per glucose) and an increased reliance on glycolysis.

Exercise training is considered the gold standard approach to enhanced cardiorespiratory fitness and peripheral insulin sensitivity across the lifespan. Metformin also benefits glycemic control and reduces cardiovascular risk. Although the evidence is not conclusive, metformin has been shown to potentially decrease exercise capacity in healthy subjects and those with metabolic syndrome. Importantly, due to the increased reliance on anaerobic metabolism, metformin may reduce the lactate threshold (LT) and lactate turn point (LTP), which are strong predictors of perception of effort, submaximal fitness, and endurance performance. Given cardiorespiratory fitness, strength, glucose control, and insulin sensitivity are predictors of disease, disability, and all-cause mortality, it is important to determine the effects of metformin on cardiorespiratory fitness and physical function.

While these mechanisms of metformin in skeletal muscle are compelling for glucose regulation, there is significant variation in the literature on the effects of metformin on exercise capacity, largely due to differences in dosing (e.g., ~50-500 mg/kg) and exercise intervention design (e.g., acute vs. short-term or chronic exercise and/or submaximal vs. maximal exercise intensity). A recent meta-analysis by found that because previous studies have predominantly used exercise intensities well below VO2max, metformin does not appear to affect maximal oxygen uptake in healthy volunteers; metformin may only alter exercise capacity at high or near-maximal work rates. Thus, there is a lack of data on the effects of metformin on lactate threshold, blood lactate clearance, and exercise-induced fatigue.

Data from this study will provide valuable insight into the effects of metformin compared to placebo on exercise capacity at near-maximal work rates in young, healthy adults. While some studies have examined metformin's impact on exercise performance, these tend to be studies where exercise intensity was well below maximal effort, in highly trained cyclists, or in clinical populations (e.g., individuals with T2DM). Importantly, the results from this study may lead healthy individuals to adjust exercise protocols to accommodate for the decline in performance along with an increased perceived exertion that may accompany metformin consumption. Moreover, this study may fill the gap in literature on a slightly longer timeline for metformin ingestion effects on exercise capacity compared to acute consumption, which may have a more profound impact on cardiorespiratory fitness and capacity over time.

ELIGIBILITY:
Inclusion Criteria:

* 18-30 years old
* Metformin-naïve
* BMI < 30 kg/m2
* Recreationally active (≥ 3 days/week of exercise)
* Females must be premenopausal and report normal menstrual cycles
* Willingness and ability to comply with scheduled visits and study procedures.

Exclusion Criteria:

* History of cardiometabolic disease, such as type 1 or type 2 diabetes
* Smoking (must have quit at least 6 mos prior)
* Use of medication that significantly alters glucose regulation (e.g., metformin, insulin, GLP-1 receptor agonists, SGLT-2 inhibitors, biguanides)
* Severe liver or kidney disease, or medications to treat liver or kidney disease
* Pregnant, breastfeeding, or plans to become pregnant during study period

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Estimated)
Dates: Start 2025-01-31 (Actual); Primary Completion 2026-04-01 (Estimated); Study Completion 2026-04-01 (Estimated)

PRIMARY OUTCOMES:
Exercise capacity | 6 weeks
  Exercise capacity will be measured by absolute and relative VO2peak
Lactate threshold | 6 weeks
  Lactate threshold (LT) will be determined by power output immediately before the curvilinear increase in lactate concentration
VO2 at Lactate threshold | 6 weeks
  VO2 at LT denoted as VO2 obtained at the same power output as LT
Lactate turnpoint (LTP) | 6 weeks
  LTP will be determined by the power output obtained immediately before the second sharp increase in blood lactate concentration
Maximal power output | 6 weeks
  Maximal power output (watts) during exercise

SECONDARY OUTCOMES:
Respiratory exchange ratio (RER) | 6 weeks
  RER will be determined during exercise as the ratio of expired CO2 and inspired O2, as an estimate of substrate utilization
Ventilation (VE) | 6 weeks
  Minute ventilation collected during exercise
Maximal fat oxidation (Fatmax) | 6 weeks
  Maximal amount of fat oxidized during exercise

OTHER OUTCOMES:
Resting blood pressure | 6 weeks
  Blood pressure obtained before exercise in a resting state
Blood pressure during exercise | 6 weeks
  Blood pressure measured during exercise at end of each stage
Resting heart rate | 6 weeks
  Heart rate obtained before exercise in a resting state
Heart rate during exercise | 6 weeks
  Heart rate measured during exercise at end of each stage
Rating of perceived exertion (RPE) | 6 weeks
  Participant-perceived difficulty of exercise recorded at end of each stage during exercise

CONTACTS AND LOCATIONS:
Overall Officials: Jason D Allen, PhD, Principal Investigator — University of Virginia
Locations (1):
- University of Virginia, Charlottesville, Virginia, United States

IPD SHARING:
Plan to Share IPD: No